CLINICAL TRIAL: NCT06585033
Title: Spinal Cord Stimulation for the Treatment of Therapy-Resistant Neuropathic Pain After Lumbar Spinal Surgery - A Randomized, Double-Blind, Sham-Controlled, Cross-over Study
Brief Title: Placebo Effect In Spinal Cord Electrical Stimulation for Pain
Acronym: PISCES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Kliment Gatzinsky, MD, PhD, Associate Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PISCES study
Record Dates: First submitted 2024-09-02; First posted 2024-09-05 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Chronic Postoperative Pain
Keywords: Spinal cord stimulation; Lumbar spine surgery; Chronic pain; Pain reduction; Placebo; Randomized controlled trial
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No stimulation (Sham Comparator)
  Interventions: Device: Spinal cord stimulation
- Stimulation (Active Comparator)
  Interventions: Device: Spinal cord stimulation

INTERVENTIONS:
Device: Spinal cord stimulation — Stimulation off
  Arms: No stimulation
Device: Spinal cord stimulation — Stimulation on
  Arms: Stimulation

SUMMARY:
Objective: To evaluate if spinal cord stimulation (SCS) performs better than placebo (no stimulation) in the long term to reduce persistent neuropathic leg pain refractory to medication and other conservative treatments in patients who have undergone lumbar spinal surgery.

Study design: Multicenter, double blind, randomized, sham-controlled trial.

After a positive SCS test trial, participants (18-70 years) will be implanted with a non-rechargeable SCS system providing active, subthreshold stimulation and followed for 12 months in a blinded cross-over design. The primary outcome measure is the difference in change in leg pain intensity scores using the Numeric Rating Scale (NRS) between a 3-month period with optimized subthreshold stimulation, and a 3-month period with no stimulation, as compared to baseline. Quality of life, physical functioning, sleep quality, return to work, and reduction in medication use will also be investigated.

Background: Up to 20% of patients who have undergone lumbar spinal surgery experience persistent back/leg pain leading to long-term reduction in functionality and quality of life. SCS is an established and safe, minimally invasive treatment for these patients when no further surgery is indicated and conservative therapies have been found to be ineffective. Placebo-controlled studies, comparing active and sham stimulation, were lacking until recently as traditional SCS relied on the patient feeling the stimulation (paresthesia). Technological progress with development of paresthesia-free stimulation forms now allows for the execution of placebo-controlled studies. A recent trial showing no significant difference in long-term effectiveness between active SCS and sham suffers from significant methodological shortcomings. This necessitates further sham-controlled studies to determine the effectiveness of SCS.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE

   SCS is an established and safe, minimally invasive treatment for patients with therapy-resistant chronic neuropathic pain. The treatment is based on the development of the gate-control theory presented in the mid-1960s as a way to dampen pain impulses at the spinal cord level. SCS treatment involves the insertion of electrode(s) in the epidural space, delivering weak electrical stimulation to the dorsal columns of the spinal cord to block pain impulses traveling to the brain. In patients experiencing sufficient pain relief (usually pain reduction over 50%) during a test trial period, an implantable pulse generator (IPG) is placed under the skin and connected to the electrode(s). Patients with chronic neuropathic pain may experience pain relief with SCS when other more invasive, surgical, and conservative treatments have been attempted and appeared to be ineffective.

   The most common condition treated with SCS is enduring neuropathic back and/or leg pain after lumbar spinal surgeries, such as lumbar discectomy. Up to 20% of patients who have undergone lumbar spinal surgery for degenerative conditions exhibit new or persistent low back/leg pain, leading to impaired functionality and reduced quality of life. This condition is entitled persistent spinal pain syndrome type 2 (PSPS2, formerly known as failed back surgery syndrome). Randomized controlled trials (RCTs) with SCS have shown long-term pain reduction of up to 70-80% in this patient group. In these studies, the effectiveness of SCS is based on either comparing different forms of stimulation or comparing SCS with reoperations and medication treatments. However, placebo/sham-controlled studies, comparing active stimulation with inactive stimulation, were lacking until recently since traditional SCS relied on the patient feeling the stimulation (paresthesia), making it impossible to conduct blinded studies where the patient does not know if the stimulation is on or off. This has constituted a major disadvantage in terms of the strength of the scientific evidence for the effect of SCS treatment, as it is known that the placebo effect is significant in surgical treatments.

   New SCS treatments for pain in which the patient does no longer experience paresthesia have been developed in recent years, which allows the execution of sham-controlled studies. A recently published study showed no significant difference between SCS and sham stimulation in long-term pain relief and improving physical functioning in patients with PSPS2, raising doubts about the effectiveness and use of the treatment, which is costly due to high material costs. However, this single study has significant methodological shortcomings. This necessitates further sham-controlled studies to ascertain whether SCS is an adequate treatment for chronic pain. The aim of the current study is to compare the long-term effect of paresthesia-free SCS with a sham treatment (no stimulation) in reducing neuropathic pain in patients with PSPS2. It is hypothesized that SCS treatment will be superior compared to treatment with sham stimulation.
2. OBJECTIVES

   Primary Objective: To compare active subthreshold SCS with sham stimulation in reducing neuropathic leg pain.

   Secondary Objective(s): To compare subthreshold SCS with sham stimulation on:
   1. quality of life
   2. physical functioning
   3. sleep quality
   4. medication use
   5. return to work
3. STUDY DESIGN

This is an international, multicenter, double-blind, randomized, sham-controlled study. Patients evaluated as candidates for SCS will after a positive test trial be implanted with the non-rechargeable Boston Alpha Prime system (Boston Sci, Marlborough, MA, USA) providing active subthreshold stimulation forms that the patient does not feel (i.e., paresthesia-free) and are proven to be effective in reducing chronic neuropathic pain. According to standard clinical practice, research participants are implanted with electrode(s) during an initial surgery, which are inserted into the epidural space posterior to the spinal cord dorsal columns, with the aim of obtaining the best possible coverage of the painful area. Subsequently, patients undergo a trial phase of 2 weeks with an external IPG to determine if treatment with a subthreshold stimulation provides adequate pain relief (over 50% pain reduction). If no adequate pain relief is experienced during the trial phase, the electrode(s) are removed and the patient is excluded from further study participation. In patients responding with adequate pain relief, a permanent IPG is placed under the skin and connected to the electrode(s). Patients will then be randomized into either the active subthreshold stimulation or sham stimulation group. After randomization, patients will undergo a four-week period where stimulation settings will be optimized and patients can recover from their surgery.

After the optimization period, patients will receive either subthreshold or sham stimulation in accordance with the randomization. The subthreshold stimulation form that will be used will be based on patient response in terms of optimal pain reduction during the 2-week trial and the 4-week optimization period. Patients can use any of the subthreshold stimulation forms or combinations that are available within the Alpha Prime system. After 3 months, patients will switch to the other stimulation group according to a crossover design, where they will receive the other stimulation form until the 6-month follow-up. Subsequently, patients will receive the stimulation form they found most effective for an additional 6 months until the end of the study. Both the physician who implanted the system and the patient will be unaware of the stimulation type received (a double-blind design) during the entire study period. Patients will be aware they will receive two different stimulation forms, while being unaware of the fact that one of the stimulation forms is sham stimulation. Activation/deactivation and programming of the stimulation will be performed by a research nurse, who is the only person in the study aware of which group the patient belongs to. Subjects enrolled will be asked to complete several questionnaires prior to their procedure and at routine follow up visits at 3, 6 and 12 months. After study termination at the 12-month follow-up, blinding will be lifted and patients can receive any stimulation form available within the Boston Alpha Prime system.

ELIGIBILITY:
Inclusion Criteria:

* History consistent with PSPS2 of at least 6 months after the last spinal surgery. The patient experienced no effect of conservative treatments and has been assessed as not eligible for further spinal surgery.
* Patients between 18-70 years of age.
* Average perceived pain intensity in one or both legs of 5 or more and average perceived pain intensity in the back of less than 3 measured with the validated 11-box NRS (0 no pain, 10 worst imaginable pain)
* The patient should have been informed verbally and in writing about the study and should have provided informed written consent to participate.
* Adequate pain relief effect (50% or more) after a two week trial with active test stimulation.

Exclusion Criteria:

* Subject is unable to understand or operate the SCS device.
* Subject currently has an active implantable device including pacemakers, spinal cord stimulator or intrathecal drug delivery system.
* Ongoing coagulation disorder.
* Ongoing abuse of alcohol, drugs, or prescription opioids.
* Active debilitating psychiatric illness.
* Active malignancy.
* Condition with increased general infection sensitivity, such as known immunodeficiency.
* Expected lifespan <1 year.
* Ongoing local infection or other skin disease where the IPG is planned to be placed.
* Pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison between active subthreshold spinal cord stimulation and sham stimulation in reducing neuropathic leg pain | Baseline and 3+3 months
  The difference in change in neuropathic leg pain intensity scores measured by the numeric rating scale (NRS) questionnaire using a 0-10 scale between a 3-month period with subthreshold stimulation and a 3-month period with sham stimulation, as compared to baseline. Zero means no pain and 10 means the worst pain imaginable with higher scores indicating worse outcome.

SECONDARY OUTCOMES:
Comparison between active subthreshold spinal cord stimulation and sham stimulation | Baseline and 3, 6 and 12 months
  Physical functioning measured using the Oswestry Disability Index (ODI) questionnaire with an index range of 0-100. Zero is equated with no disabiliy and 100 is the maximum disability possible with higher scores indicating a worse outcome.
Comparison between active subthreshold spinal cord stimulation and sham stimulation | Baseline and 3, 6 and 12 months
  • Quality of life measured using the EuroQoL-5 Dimension-5 Levels (EQ-5D-5L) questionnaire assigning values of 1 (no problems) to 5 (extreme problems) and summing these values cross five items, resulting in a score from 5 (no problems on any dimensions) to 25 (extreme problems on all dimensions). Higher scores mean worse outcome.
Comparison between active subthreshold spinal cord stimulation and sham stimulation | Baseline and 3, 6 and 12 months
  Sleep quality measured using the Pittsburgh Sleep Quality Index (PSQI) seven component questionnaire with each component scoring from 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0-21) where higher scores indicate worse sleep quality.
Comparison between active subthreshold spinal cord stimulation and sham stimulation | Baseline and 3, 6 and 12 months
  Medication use
Comparison between active subthreshold spinal cord stimulation and sham stimulation | Baseline and 3, 6 and 12 months
  Number of hours worked per week
Comparison between active subthreshold spinal cord stimulation and sham stimulation | Baseline and 12 months
  The difference in change in neuropathic leg pain intensity scores, compared to baseline, measured by the numeric rating scale (NRS) questionnaire using a 0-10 scale after patient has chosen the preferred stimulation from the 6-month to the 12-month follow-up. Zero means no pain and 10 means the worst pain imaginable with higher scores indicating worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kliment Gatzinsky, MD, PhD, Principal Investigator — Department of Neurosurgery, Sahlgrenska University Hospital
Locations (4):
- Department of Anaesthesiology and Pain Management, Rijnstate Hospital, Arnhem, Netherlands
- Department of Neurosurgery, Stavanger University hospital, Stavanger, Norway
- Sweden (2):
  - Department of Neurosurgery, Sahlgrenska University Hospital, Gothenburg
  - Department of Anesthesiology and Intensive Care/Pain Center, Sahlgrenska University Hospital Östra, Gothenburg

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported, after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Deer TR, Mekhail N, Provenzano D, Pope J, Krames E, Leong M, Levy RM, Abejon D, Buchser E, Burton A, Buvanendran A, Candido K, Caraway D, Cousins M, DeJongste M, Diwan S, Eldabe S, Gatzinsky K, Foreman RD, Hayek S, Kim P, Kinfe T, Kloth D, Kumar K, Rizvi S, Lad SP, Liem L, Linderoth B, Mackey S, McDowell G, McRoberts P, Poree L, Prager J, Raso L, Rauck R, Russo M, Simpson B, Slavin K, Staats P, Stanton-Hicks M, Verrills P, Wellington J, Williams K, North R; Neuromodulation Appropriateness Consensus Committee. The appropriate use of neurostimulation of the spinal cord and peripheral nervous system for the treatment of chronic pain and ischemic diseases: the Neuromodulation Appropriateness Consensus Committee. Neuromodulation. 2014 Aug;17(6):515-50; discussion 550. doi: 10.1111/ner.12208. PMID 25112889
- [Background] Gatzinsky K. Spinal cord stimulation. In: Knotkova H, Rasche D, eds. Textbook of Neuromodulation: Principles, Methods and Clinical Applications. New York: Springer; 2015:35-52.
- [Background] Zheng Y, Liu CW, Hui Chan DX, Kai Ong DW, Xin Ker JR, Ng WH, Wan KR. Neurostimulation for Chronic Pain: A Systematic Review of High-Quality Randomized Controlled Trials With Long-Term Follow-Up. Neuromodulation. 2023 Oct;26(7):1276-1294. doi: 10.1016/j.neurom.2023.05.003. Epub 2023 Jul 10. PMID 37436342
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Amirdelfan K, Webster L, Poree L, Sukul V, McRoberts P. Treatment Options for Failed Back Surgery Syndrome Patients With Refractory Chronic Pain: An Evidence Based Approach. Spine (Phila Pa 1976). 2017 Jul 15;42 Suppl 14:S41-S52. doi: 10.1097/BRS.0000000000002217. PMID 28505029
- [Background] Rigoard P, Gatzinsky K, Deneuville JP, Duyvendak W, Naiditch N, Van Buyten JP, Eldabe S. Optimizing the Management and Outcomes of Failed Back Surgery Syndrome: A Consensus Statement on Definition and Outlines for Patient Assessment. Pain Res Manag. 2019 Feb 18;2019:3126464. doi: 10.1155/2019/3126464. eCollection 2019. PMID 30911339
- [Background] Gatzinsky K, Eldabe S, Deneuville JP, Duyvendak W, Naiditch N, Van Buyten JP, Rigoard P. Optimizing the Management and Outcomes of Failed Back Surgery Syndrome: A Proposal of a Standardized Multidisciplinary Team Care Pathway. Pain Res Manag. 2019 Jul 8;2019:8184592. doi: 10.1155/2019/8184592. eCollection 2019. PMID 31360272
- [Background] Parker SL, Mendenhall SK, Godil SS, Sivasubramanian P, Cahill K, Ziewacz J, McGirt MJ. Incidence of Low Back Pain After Lumbar Discectomy for Herniated Disc and Its Effect on Patient-reported Outcomes. Clin Orthop Relat Res. 2015 Jun;473(6):1988-99. doi: 10.1007/s11999-015-4193-1. PMID 25694267
- [Background] Weir S, Samnaliev M, Kuo TC, Ni Choitir C, Tierney TS, Cumming D, Bruce J, Manca A, Taylor RS, Eldabe S. The incidence and healthcare costs of persistent postoperative pain following lumbar spine surgery in the UK: a cohort study using the Clinical Practice Research Datalink (CPRD) and Hospital Episode Statistics (HES). BMJ Open. 2017 Sep 11;7(9):e017585. doi: 10.1136/bmjopen-2017-017585. PMID 28893756
- [Background] Kapural L, Yu C, Doust MW, Gliner BE, Vallejo R, Sitzman BT, Amirdelfan K, Morgan DM, Brown LL, Yearwood TL, Bundschu R, Burton AW, Yang T, Benyamin R, Burgher AH. Novel 10-kHz High-frequency Therapy (HF10 Therapy) Is Superior to Traditional Low-frequency Spinal Cord Stimulation for the Treatment of Chronic Back and Leg Pain: The SENZA-RCT Randomized Controlled Trial. Anesthesiology. 2015 Oct;123(4):851-60. doi: 10.1097/ALN.0000000000000774. PMID 26218762
- [Background] Veizi E, Hayek SM, North J, Brent Chafin T, Yearwood TL, Raso L, Frey R, Cairns K, Berg A, Brendel J, Haider N, McCarty M, Vucetic H, Sherman A, Chen L, Mekel-Bobrov N. Spinal Cord Stimulation (SCS) with Anatomically Guided (3D) Neural Targeting Shows Superior Chronic Axial Low Back Pain Relief Compared to Traditional SCS-LUMINA Study. Pain Med. 2017 Aug 1;18(8):1534-1548. doi: 10.1093/pm/pnw286. PMID 28108641
- [Background] Deer T, Slavin KV, Amirdelfan K, North RB, Burton AW, Yearwood TL, Tavel E, Staats P, Falowski S, Pope J, Justiz R, Fabi AY, Taghva A, Paicius R, Houden T, Wilson D. Success Using Neuromodulation With BURST (SUNBURST) Study: Results From a Prospective, Randomized Controlled Trial Using a Novel Burst Waveform. Neuromodulation. 2018 Jan;21(1):56-66. doi: 10.1111/ner.12698. Epub 2017 Sep 29. PMID 28961366
- [Background] Mekhail N, Levy RM, Deer TR, Kapural L, Li S, Amirdelfan K, Hunter CW, Rosen SM, Costandi SJ, Falowski SM, Burgher AH, Pope JE, Gilmore CA, Qureshi FA, Staats PS, Scowcroft J, Carlson J, Kim CK, Yang MI, Stauss T, Poree L; Evoke Study Group. Long-term safety and efficacy of closed-loop spinal cord stimulation to treat chronic back and leg pain (Evoke): a double-blind, randomised, controlled trial. Lancet Neurol. 2020 Feb;19(2):123-134. doi: 10.1016/S1474-4422(19)30414-4. Epub 2019 Dec 20. PMID 31870766
- [Background] North RB, Kidd DH, Farrokhi F, Piantadosi SA. Spinal cord stimulation versus repeated lumbosacral spine surgery for chronic pain: a randomized, controlled trial. Neurosurgery. 2005;56(1):98-106; discussion 106-7. doi: 10.1227/01.neu.0000144839.65524.e0. PMID 15617591
- [Background] Kumar K, Taylor RS, Jacques L, Eldabe S, Meglio M, Molet J, Thomson S, O'Callaghan J, Eisenberg E, Milbouw G, Buchser E, Fortini G, Richardson J, North RB. Spinal cord stimulation versus conventional medical management for neuropathic pain: a multicentre randomised controlled trial in patients with failed back surgery syndrome. Pain. 2007 Nov;132(1-2):179-88. doi: 10.1016/j.pain.2007.07.028. Epub 2007 Sep 12. PMID 17845835
- [Background] Deer T, Gilligan C, Falowski S, Desai M, Pilitsis J, Jameson J, Moeschler S, Heros R, Tavel E, Christopher A, Patterson D, Wahezi S, Weisbein J, Antony A, Funk R, Ibrahim M, Lim C, Wilson D, Fishell M, Scarfo K, Dickerson D, Braun E, Buchanan P, Levy RM, Miller N, Duncan J, Xu J, Candido K, Kreiner S, Fahey ME, Yue J. Treatment of Refractory Low Back Pain Using Passive Recharge Burst in Patients Without Options for Corrective Surgery: Findings and Results From the DISTINCT Study, a Prospective Randomized Multicenter Controlled Trial. Neuromodulation. 2023 Oct;26(7):1387-1399. doi: 10.1016/j.neurom.2023.07.009. Epub 2023 Aug 28. PMID 37642628
- [Background] Dettori JR, Norvell DC, Chapman JR. The Art of Surgery: The Strange World of the Placebo Response. Global Spine J. 2019 Sep;9(6):680-683. doi: 10.1177/2192568219861972. Epub 2019 Jul 17. No abstract available. PMID 31448203
- [Background] Karjalainen T, Heikkinen J, Busija L, Jokihaara J, Lewin AM, Naylor JM, Harris L, Harris IA, Buchbinder R, Adie S. Use of Placebo and Nonoperative Control Groups in Surgical Trials: A Systematic Review and Meta-analysis. JAMA Netw Open. 2022 Jul 1;5(7):e2223903. doi: 10.1001/jamanetworkopen.2022.23903. PMID 35895060
- [Background] Duarte RV, Nevitt S, McNicol E, Taylor RS, Buchser E, North RB, Eldabe S. Systematic review and meta-analysis of placebo/sham controlled randomised trials of spinal cord stimulation for neuropathic pain. Pain. 2020 Jan;161(1):24-35. doi: 10.1097/j.pain.0000000000001689. PMID 31453983
- [Background] Hara S, Andresen H, Solheim O, Carlsen SM, Sundstrom T, Lonne G, Lonne VV, Taraldsen K, Tronvik EA, Oie LR, Gulati AM, Sagberg LM, Jakola AS, Solberg TK, Nygaard OP, Salvesen OO, Gulati S. Effect of Spinal Cord Burst Stimulation vs Placebo Stimulation on Disability in Patients With Chronic Radicular Pain After Lumbar Spine Surgery: A Randomized Clinical Trial. JAMA. 2022 Oct 18;328(15):1506-1514. doi: 10.1001/jama.2022.18231. PMID 36255427
- [Background] Thomson S, Kallewaard JW, Gatzinsky K. Spinal Cord Burst Stimulation vs Placebo Stimulation for Patients With Chronic Radicular Pain After Lumbar Spine Surgery. JAMA. 2023 Mar 14;329(10):847. doi: 10.1001/jama.2022.24742. No abstract available. PMID 36917057
- [Background] Taylor RS, Eldabe S. Placebo (Sham) Controlled Trials of Spinal Cord Stimulation. Neuromodulation. 2023 Feb;26(2):474-475. doi: 10.1016/j.neurom.2022.11.013. Epub 2022 Dec 15. No abstract available. PMID 36526546
- [Background] Paz-Solis J, Thomson S, Jain R, Chen L, Huertas I, Doan Q. Exploration of High- and Low-Frequency Options for Subperception Spinal Cord Stimulation Using Neural Dosing Parameter Relationships: The HALO Study. Neuromodulation. 2022 Jan;25(1):94-102. doi: 10.1111/ner.13390. PMID 35041592
- [Background] Thomson SJ, Tavakkolizadeh M, Love-Jones S, Patel NK, Gu JW, Bains A, Doan Q, Moffitt M. Effects of Rate on Analgesia in Kilohertz Frequency Spinal Cord Stimulation: Results of the PROCO Randomized Controlled Trial. Neuromodulation. 2018 Jan;21(1):67-76. doi: 10.1111/ner.12746. Epub 2017 Dec 8. PMID 29220121
- [Background] Metzger CS, Hammond MB, Paz-Solis JF, Newton WJ, Thomson SJ, Pei Y, Jain R, Moffitt M, Annecchino L, Doan Q. A novel fast-acting sub-perception spinal cord stimulation therapy enables rapid onset of analgesia in patients with chronic pain. Expert Rev Med Devices. 2021 Mar;18(3):299-306. doi: 10.1080/17434440.2021.1890580. Epub 2021 Mar 3. PMID 33656411